CLINICAL TRIAL: NCT00560092
Title: Effects of a Single Dose of Intrathecal Magnesium Sulfate on Postoperative Morphine Consumption After Total Hip Replacement
Brief Title: Intrathecal Magnesium and Postoperative Analgesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CHU63-006
Record Dates: First submitted 2006-06-22; First posted 2007-11-19 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Total Hip Replacement
Keywords: Magnesium; Pain; Morphine; Intrathecal; NMDA; Elective total hip replacement under intrathecal anesthesia
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- intrathecal magnesium sulfate (Experimental)
  Interventions: Drug: intrathecal magnesium sulfate

INTERVENTIONS:
Drug: intrathecal magnesium sulfate — intrathecal magnesium sulfate

SUMMARY:
Magnesium is implicated in the activation of NMDA receptors by amino-excitatory acids in the central nervous system [1]. Magnesium deficiency is associated to an increased activation of these receptors, and to an increased sensitivity to pain in animals. Spinal cord is the site of sensitization of pain, mainly mediated by the NMDA receptors, and intrathecal magnesium may have anti-hyperalgesic effect when administered intrathecally [2]. As intrathecal magnesium has already been used in humans for treatment of eclampsia, we stated that it could also improve postoperative analgesia and reduce the need for auto-administered morphine if given (50 mg of magnesium sulfate) with the intrathecal anesthetic drugs (bupivacaine and sufentanil) injected for orthopedic surgery.

DETAILED DESCRIPTION:
Magnesium is implicated in the activation of NMDA receptors by amino-excitatory acids in the central nervous system [1]. Magnesium deficiency is associated to an increased activation of these receptors, and to an increased sensitivity to pain in animals. Spinal cord is the site of sensitization of pain, mainly mediated by the NMDA receptors, and intrathecal magnesium may have anti-hyperalgesic effect when administered intrathecally [2]. As intrathecal magnesium has already been used in humans for treatment of eclampsia, we stated that it could also improve postoperative analgesia and reduce the need for auto-administered morphine if given (50 mg of magnesium sulfate) with the intrathecal anesthetic drugs (bupivacaine and sufentanil) injected for orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Total hip replacement under intrathecal anesthesia.

Exclusion Criteria:

* General anesthesia (alone or not)
* Intolerance to morphine
* Misunderstanding of the use of the device for intravenous patient-controlled administration of morphine.

Ages: 56 Years to 93 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Reduction of morphine consumption in the postoperative period. | in the postoperative period

SECONDARY OUTCOMES:
Duration of sensory and motor blockade induced by the intrathecal anesthesia ; side effects; postoperative pain (visual analogue scale). | postoperative pain

CONTACTS AND LOCATIONS:
Overall Officials: Christian Duale, Dr, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Background] Mayer ML, Westbrook GL. Permeation and block of N-methyl-D-aspartic acid receptor channels by divalent cations in mouse cultured central neurones. J Physiol. 1987 Dec;394:501-27. doi: 10.1113/jphysiol.1987.sp016883. PMID 2451020
- [Background] Buvanendran A, McCarthy RJ, Kroin JS, Leong W, Perry P, Tuman KJ. Intrathecal magnesium prolongs fentanyl analgesia: a prospective, randomized, controlled trial. Anesth Analg. 2002 Sep;95(3):661-6, table of contents. doi: 10.1097/00000539-200209000-00031. PMID 12198056